CLINICAL TRIAL: NCT04748562
Title: Vaginal Progesterone 400mg v.s 200mg for Prevention of Preterm Labor in Twin Pregnancies: a Randomised Controlled Trial
Brief Title: Vaginal Progesterone 400mg v.s 200mg for Prevention of Preterm Labor in Twin Pregnancies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MS 483/2019
Record Dates: First submitted 2021-01-31; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Twin Pregnancy With Antenatal Problem
Keywords: Progesterone; Twin pregnancy; Preterm labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 400 mg progesterone group (Active Comparator): Taking 400 mg vaginal progesterone
  Interventions: Drug: Progesterone
- 200 mg progesterone group (Active Comparator): Taking 200 mg vaginal progesterone
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — Taking prontogest vaginally

SUMMARY:
It is already known that the risk of preterm labor in twin pregnancy before 37 week is 8-9 fold higher compared to singletons, and progesterone supplementation can decrease the incidence of preterm labor in singleton pregnancy.

There were studies that used 200mg vaginal progesterone with no effect on the result So this study aims To examine the effect of prophylactic vaginal progesterone 400mg v.s 200mg for prevention of preterm birth in twin pregnancies

ELIGIBILITY:
Inclusion Criteria:

1. Primigravidae
2. Twin pregnancies at gestational age 14 week.
3. Cervical length more than 2 cm (because if 2cm or less they will undergo cervical cerclage.)

Exclusion Criteria:

* Polyhydramnios
* Anemia
* Twins with congenital malformation
* Twin to twin transfusion
* Medical diseases as diabetes mellitus, hypertension and systemic lupus erythematosis
* Previous cervical surgery
* High order pregnancy (triples or more)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Preterm labor | Before 37 weeks gestation
  Number of participants which had preterm labor

SECONDARY OUTCOMES:
Cervical length changes | Between 14 weeks and 22 weeks gestation
  Cervical length changes in centimeters
Neonatal ICU admission | The first 28 days after delivery
  Number of neonates required neonatal ICU admission
Neonatal mechanical ventilation | The first 28 days after delivery
  Number of neonates required mechanical ventilation
Progesterone side effects | During one year which is the period from the start of the study till its end
  The number of patients experiencing progesterone side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided